CLINICAL TRIAL: NCT01441609
Title: Effect of the Expression Level of Th9 Cells and IL-9 In Poor/Non-responsiveness to Hepatitis B Vaccination
Brief Title: Expression of Th9 Cells and Poor/Non-responsiveness to Hepatitis B Vaccination
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Principal Investigator, Wu Jiang, Director, Centers for Disease Control and Prevention
Other Study IDs: BJCDCWJ201103
Record Dates: First submitted 2011-09-26; First posted 2011-09-27 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Hepatitis B
Keywords: Th9 cells; IL9; non/poor responsiveness to hepatitis B; collect blood samples after vaccination
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- the value of anti-HBs =0 mIU/ml: Recent serological testing result show HBsAg, HBeAg, anti-HBe, anti-HBc, HBV DNA and Pre-S1 should be negative. had vaccinated hepatitis B vaccine and the value of anti-HBs be zero.
- the value of anti-HBs≤5mIU/ml: Recent serological testing result show HBsAg, HBeAg, anti-HBe, anti-HBc, HBV DNA and Pre-S1 should be negative. had vaccinated hepatitis B vaccine and the value of anti-HBs≤5mIU/ml.
- 5mIU≤anti-HBs≤10mIU/ml: Recent serological testing result show HBsAg, HBeAg, anti-HBe, anti-HBc, HBV DNA and Pre-S1 should be negative. had vaccinated hepatitis B vaccine and the value of 5mIU≤anti-HBs≤10mIU
- anti-HBs≥1000mIU: Recent serological testing result show HBsAg, HBeAg, anti-HBe, anti-HBc, HBV DNA and Pre-S1 should be negative. had vaccinated hepatitis B vaccine and the value of anti-HBs≥1000mIU.

SUMMARY:
An observational study will be performed in subjects aged 3-65 years old to describe the dynamic changes of cellular immunity after vaccination of hepatitis B vaccine, and to find out the expression levels of Th9 cells and IL9 in subjects with different response to the primary immunization (3 single -dose injunctions).

DETAILED DESCRIPTION:
This study selected 74 volunteers which had the hepatitis B vaccine (immunization programs 0,1,6) , anti-HBs≤10mIU as the research subjects, and choose 20 volunteers which anti-HBs≥1000mIU as the control group, revaccination the groups according to the normal immunization programs, then the blood samples would be collected at 7th day, separate the PBMC and detect the expression levels of Th9 cells and IL9 by FCM, trying to find out the effects of Th9 and IL9 of non/poor -responsiveness subjects to hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* volunteer
* between 3-60 years old
* healthy
* have the history of vaccination of hepatitis B.
* Recent serological testing result show HBsAg, HBeAg, anti-HBe, anti-HBc, HBV DNA and Pre-S1 should be negative.
* informed consent
* not allergic to the component of the vaccine

Exclusion Criteria:

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 94 subjects divided into 4 groups
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-04 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Th9 cells | blood sample of 7th day after each vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Wu Jiang, Study Director — main investigator
Locations (1):
- Chifeng, Inner Mongolia, China